CLINICAL TRIAL: NCT05738577
Title: Apelin as a Marker of Early Complications in Type 1 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reem Mostafa Mohamed Sholkamy, resident doctor, Assiut University
Other Study IDs: assiut123
Record Dates: First submitted 2023-01-12; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Apelin
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: patients with type 1 diabetes aged 20-30 years
- 2: healthy people serve as controls of the same age group

SUMMARY:
Aims of the Research :

1. assessment of serum apelin levels in patients with T1DM with comparison to non-diabetic controls.
2. investigate the relation between serum apelin levels and glycemic balance.
3. clarify the the relation between serum apelin and lipid concentrations.

DETAILED DESCRIPTION:
Type 1 Diabetes Mellitus (T1DM) is an endocrine disorder in which pancreatic β cells stop producing insulin due to autoimmune destruction. This results in hyperglycemia and ketosis ; thus insulin replacement is vital in management . Incidence peaks in puberty and early adulthood . Symptoms include polyuria , polydepsia and weight loss. T1DM can cause micro and macrovascular complications which affect the quality of life .

.Studies proved that TIDM is associated with metabolic abnormalities and alteration of adipose tissue hormones (adipokines). Adipose tissue yields many adipocytokines that modulate insulin sensitivity and play essential role in the pathogenesis of diabetes . Given these complications, we strive to discover new targets that enable us to control DM. One of these targets is apelin .

Apelin is an adipocytokine widely distributed throughout the body including skeletal muscle, cardiac muscle, pulmonary tissue, mammary glands, ovaries, brain, kidneys, pancreas and adrenal glands.It was extracted from the bovine stomach by Tatemoto et al., in 1998.

Apelin plays a role in a range of physiological processes including regulation of fluid hemostasis and blood pressure ,improvement of cardiac contractility ,lipid metabolism and metabolic control. It appears to improve insulin sensitivity, reduces blood glucose and increases glucose utilisation .

It has been shown that apelin has a crucial role in energy metabolism and pathogenesis of diabetes mellitus and its level is altered in diabetic patients .High serum apelin level was linked to impaired insulin sensitivity . Thus, it was suggested that serum apelin can be used for the prediction of development of diabetes and its progression .

Serum cholesterol, triglycerides (TG) and LDL are significantly increased in T1DM, but serum HDL is decreased . So, patients with T1DM are at high risk of developing premature atherosclerosis because of hyperlipidemia. A correlation was found between serum apelin and cholesterol, TG and LDL in diabetic patients .

. Apelin was shown to increase the stability of lipid vacuoles making them more resistant to lipolysis. So apelin can be used as a predictor of premature atherosclerosis in T1DM .

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetic patients (treated with insulin ). age between 20 to 30 years , including males and females.

And accepting participation in the study.

Exclusion Criteria:

* patients with acute illness.and pregnancy.

Ages: 20 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: 60 patients with Type 1 Diabetes Mellitus and 30 healthy individuals of the same age group serve as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-02-25 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
glycemic control according to apelin level | baseline

SECONDARY OUTCOMES:
Detection of the relation of apelin and lipid profile in diabetic patients | baseline

REFERENCES:
- [Background] Al-Selwi Y, Shaw JA, Kattner N. Understanding the Pancreatic Islet Microenvironment in Cystic Fibrosis and the Extrinsic Pathways Leading to Cystic Fibrosis Related Diabetes. Clin Med Insights Endocrinol Diabetes. 2021 Oct 12;14:11795514211048813. doi: 10.1177/11795514211048813. eCollection 2021. PMID 34675737
- [Background] Sabry RN, El Wakeel MA, El-Kassas GM, Amer AF, El Batal WH, El-Zayat SR, Abou-El-Asrar M. Serum Apelin: A New Marker of Early Atherosclerosis in Children with Type 1 Diabetes Mellitus. Open Access Maced J Med Sci. 2018 Apr 4;6(4):613-617. doi: 10.3889/oamjms.2018.144. eCollection 2018 Apr 15. PMID 29731925
- See also: https://dx.doi.org/10.21608/ejhm.2022.246905 — https://dx.doi.org/10.21608/ejhm.2022.246905
- See also: https://doi.org/10.1590/2359-3997000000271 — https://doi.org/10.1590/2359-3997000000271
- See also: https://doi.org/10.4103%2Fjrms.JRMS_675_20 — https://doi.org/10.4103%2Fjrms.JRMS_675_20